CLINICAL TRIAL: NCT04499794
Title: The Study of Exosome EML4-ALK Fusion in NSCLC Clinical Diagnosis and Dynamic Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yutao Liu, Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC2064
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Untreated Advanced NSCLC Patients; FISH Identified ALK Fusion Positive or Negative
MeSH Terms: interventions — 1,1'-(4,4'-(((5-chloropyrimidine-2,4-diyl)bis(azanediyl))bis(3-methoxy-4,1-phenylene))bis(piperazine-4,1-diyl))diethanone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FISH diagnosed EML4-ALK fusion positive NSCLC group
  Interventions: Drug: ALK inhibitor
- FISH diagnosed EML4-ALK fusion negative NSCLC group

INTERVENTIONS:
Drug: ALK inhibitor — ALK inhibitor treatment on ALK fusion positive NSCLC patients
  Groups: FISH diagnosed EML4-ALK fusion positive NSCLC group

SUMMARY:
The application of ALK inhibitors in the first-line cancer treatment can significantly increase the PFS and ORR of patients those with EML4-ALK fusion. The contemporary clinical ALK fusion detection are mainly via FISH and ICH while biopsies are needed. For locations where are difficult to take biopsies, these routine examinations can hardly been adopted. Apart from these, part of ALK fusion patients are resistant to ALK inhibitors, also making an accurate and efficient prognostic indicator for efficacy evaluation and identifying high-risk recurrent population an urgent priority.

The bilayer membrane structure of exosome helps maintain its internal genetic stability, making detection of EML4-ALK fusion via plasma exosomes in advanced NSCLC patients a feasible way, which might provide a non-invasive and more convenient approach for NSCLC diagnosis and efficacy monitoring. Firstly, this study will evaluate the performance of exosome EML4-ALK fusion detection in NSCLC diagnosis, which sensitivity and specificity would be compared with the FDA approved IHC (ALK [D5F3] CDx Assay) test. Subsequently, this study would monitor the dynamic changes of EML4-ALK fusion in exosome examination diagnosed ALK fusion positive NSCLC patients both before and after treatment. It aims to prospectively evaluate the potential value of this approach on efficacy and prognosis prediction in NSCLC therapy and determining whether exosome ALK fusion could assess the curative effect more accurately than imaging examination and tumor markers. Thirdly, FISH diagnosed EML4-ALK positive NSCLC patients will be divided into the positive or negative subgroup according to their post-treatment exosome ALK fusion expression which were determined at 2-3 months after ALK inhibitor were adopted. The prognostic value of monitoring exosome EML4-ALK fusion expression is assessed through the comparison of patients PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

* All eligible patients must have histologically or cytologically confirmed stage IIIB-IV unresectable NSCLC positive or negative for EML4-ALK4 fusion as defined by FISH. Patients must have an ECOG PS of 0- 1 and have at least 1 measurable lesions (RECIST 1.1 standard). For eligible patients, prior ALK inhibitor therapy or previous systemic anticancer therapy is not allowed or has been completed over 12 months. Patients with brain metastasis are eligible only in a stable central nervous system condition and treatment outcome, cannot receive glucocorticoids and drugs prohibited in the exclusion criteria ≤14 days before the first dose of study drug.

Exclusion Criteria:

* Eligible patients must not have received any major surgery ≤28 days before the first dose of study drug and must not have received any minor surgery or radiotherapy ≤14 days before the first dose of study drug. Any acute toxic reaction must have recovered to ≤ Grade 1 (except for hair loss). Patients with carcinomatous meningitis, leptomeningeal disease or spinal cord compression must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced NSCLC patients
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 6-8 weeks
  the ORR of those NSCLC patients receive ALK inhibitors treatment according to exosome ALK fusion diagnosis and FISH examination

SECONDARY OUTCOMES:
PFS | 36 months
  the PFS of those NSCLC patients receive ALK inhibitors treatment according to exosome ALK fusion diagnosis and FISH examination

CONTACTS AND LOCATIONS:
Overall Officials: Yutao LIU, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hyun KA, Kim J, Gwak H, Jung HI. Isolation and enrichment of circulating biomarkers for cancer screening, detection, and diagnostics. Analyst. 2016 Jan 21;141(2):382-92. doi: 10.1039/c5an01762a. PMID 26588824
- [Background] Cazzoli R, Buttitta F, Di Nicola M, Malatesta S, Marchetti A, Rom WN, Pass HI. microRNAs derived from circulating exosomes as noninvasive biomarkers for screening and diagnosing lung cancer. J Thorac Oncol. 2013 Sep;8(9):1156-62. doi: 10.1097/JTO.0b013e318299ac32. PMID 23945385
- [Background] Castellanos-Rizaldos E, Zhang X, Tadigotla VR, Grimm DG, Karlovich C, Raez LE, Skog JK. Exosome-based detection of activating and resistance EGFR mutations from plasma of non-small cell lung cancer patients. Oncotarget. 2019 Apr 23;10(30):2911-2920. doi: 10.18632/oncotarget.26885. eCollection 2019 Apr 23. PMID 31080561
- [Background] Tong Y, Zhao Z, Liu B, Bao A, Zheng H, Gu J, McGrath M, Xia Y, Tan B, Song C, Li Y. 5'/ 3' imbalance strategy to detect ALK fusion genes in circulating tumor RNA from patients with non-small cell lung cancer. J Exp Clin Cancer Res. 2018 Mar 27;37(1):68. doi: 10.1186/s13046-018-0735-1. PMID 29587818